CLINICAL TRIAL: NCT02304276
Title: 18F-Fluoride Assessment of Aortic Bioprosthesis Durability and Outcome
Acronym: 18F-FAABULOUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Cambridge University Hospitals NHS Foundation Trust (Other); Papworth Hospital NHS Foundation Trust (Other Government); Bichat Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 147780
Record Dates: First submitted 2014-11-10; First posted 2014-12-01 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Heart; Complications, Valve, Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Explanted valves) (Active Comparator): 10 subjects who are due to undergo repeat aortic valve replacement surgery
  Investigations:
  1. Baseline 18F-Fluoride PET-CT scan
  2. Retrieval of explanted bioprosthetic aortic valve at time of surgery for analysis
  Interventions: Radiation: 18F-Fluoride PET-CT
- 2 (AVR) (Experimental): 70 subjects with surgical bioprosthetic AVR, to include 10 subjects who have had a valve replacement < 1 month; 20 at 2 years; 20 at 5 years and 20 at >10 years.
  Investigations:
  1. Baseline 18F-Fluoride PET-CT scan
  2. Repeat CT calcium score of aortic valve at 2 years
  3. Annual clinical follow-up for 5 years (history, examination, blood tests, ECG and echocardiogram)
  Interventions: Radiation: 18F-Fluoride PET-CT; Radiation: CT calcium score of aortic valve
- 3 (TAVI) (Experimental): 50 subjects who have undergone TAVI with the COREVALVE and 50 subjects with the SAPIEN valve. In each group this will include 10 subjects who have had TAVI < 1 month; 20 at 2 years and 20 at 5 years.
  Investigations:
  1. Baseline 18F-Fluoride PET-CT scan
  2. Repeat CT calcium score of aortic valve at 2 years
  3. Annual clinical follow-up for 5 years (history, examination, blood tests, ECG and echocardiogram)
  Interventions: Radiation: 18F-Fluoride PET-CT; Radiation: CT calcium score of aortic valve

INTERVENTIONS:
Radiation: 18F-Fluoride PET-CT — Injection of 18F-Fluoride with target activity 125MBq giving an anticipated radiation exposure of 3mSv CT scanning protocol giving an anticipated radiation exposure of 13mSv
Radiation: CT calcium score of aortic valve — CT associated with an anticipated radiation exposure of 3mSv (Cohorts 2 and 3 only)
  Arms: 2 (AVR); 3 (TAVI)

SUMMARY:
This study will evaluate the two main types of replacement tissue heart valve used in current practice, comparing outcomes from surgical aortic valve replacement (AVR) with that of the more recently introduced "key-hole" procedure called transcatheter aortic valve implantation (TAVI). Participants will be recruited at various time points ranging from 1 month to 10 years following valve replacement with either AVR or TAVI. It is thought that progressive calcium (chalk) formation is responsible for the failure of the majority of these valves. All participants will therefore have a PET-CT scan with a special type of "tracer" called 18F-fluoride in order to measure active calcium formation in the valve. They will then have annual clinical follow-up for 5 years and be invited back for a repeat CT scan at 2 years to measure change in calcium burden. This study aims to investigate, firstly, the effects of valve age and type on calcium formation as measured by PET-CT and, secondly, whether this measure of calcium formation can help to predict how long different types of valve will last. If successful, 18F-fluoride PET-CT could become a valuable tool for testing new treatments to improve valve longevity and new valve designs.

DETAILED DESCRIPTION:
Aortic stenosis is the commonest form of valve disease in the western world and the leading indication for valve surgery. Bioprosthetic valves are known to degenerate via a process that is predominantly driven by calcification. Transcatheter aortic valve implantation (TAVI) has recently emerged as a less invasive alternative to conventional aortic valve replacement (AVR) surgery. Whilst this technique holds great promise, long-term follow up data are lacking and the longevity of these valves remains to be established.

In this longitudinal, cross-sectional study of 180 subjects with either surgical or transcatheter implanted bioprostheses, this study proposes to look for the earliest signs of active calcification using 18F-fluoride positron emission tomography (PET). During a 5 year follow-up period, this study hopes to demonstrate that 18F-fluoride PET will predict subsequent bioprosthetic valve degeneration and identify patients at risk of premature valve failure. The study also hopes that it will inform about the comparative durability of novel percutaneous valves. If successful, 18F-Fluoride could provide a useful method of assessing novel therapeutic strategies targeted at improving the longevity of bioprostheses and help to guide future valve design.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* able to provide informed consent
* aged over 40 years
* patients with a bioprosthetic aortic valve who are due to undergo a redo-surgical aortic valve replacement

Cohort 2

* able to provide informed consent
* aged over 40 years
* patients at 1 month (n=10), 2 years (n=20), 5 years (n=20) and 10 years (n=20) following surgical bioprosthetic aortic valve replacement

Cohort 3

* able to provide informed consent
* aged over 40 years
* patients at 1 month (n=10), 2 years (n=20) and 5 years (n=20) following transcatheter aortic valve implantation (TAVI) with the Edward's SAPIEN and the COREVALVE.

Exclusion Criteria:

* Inability to give informed consent
* Pregnancy
* Breastfeeding
* Claustrophobia
* Allergy to iodinated contrast
* Liver failure
* Chronic kidney disease (with estimated glomerular filtration rate <30 mL/min)
* Metastatic malignancy
* Paget's disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
18F-Fluoride uptake in aortic bioprostheses | Baseline
  18F-Fluoride uptake expressed as tissue to background ratio (TBR) in aortic valve bioprostheses of different age and type as measured by PET/CT

SECONDARY OUTCOMES:
CT calcium score of aortic valve | Baseline and 2 years
  Change in aortic valve calcium score (Agatston units) from baseline to 2 years as determined by CT
Echocardiographic evaluation of aortic valve function | Baseline, 1 year and 2 years
  Change in echocardiographic parameters of aortic valve function (both stenosis and regurgitation) from baseline to 1 year and 2 years as determined by Doppler echocardiography
Frequency of major adverse cardiovascular events | 5 years
  Frequency of major adverse cardiovascular events (cardiovascular death, myocardial infarction, stroke, admission with heart failure, repeat valve surgery) as determined by annual clinical follow-up of study population over 5 years
Immunohistochemical staining of explanted aortic bioprostheses for marker of calcification | intraoperative
  Immunohistochemical staining for markers of mineralisation (alkaline phosphatase, Runx-2, osteocalcin) in explanted aortic valve bioprostheses expressed as a percentage of total valve surface area.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dweck, MBChB PhD, Principal Investigator — University of Edinburgh, Scotland

REFERENCES:
- [Result] Cartlidge TRG, Doris MK, Sellers SL, Pawade TA, White AC, Pessotto R, Kwiecinski J, Fletcher A, Alcaide C, Lucatelli C, Densem C, Rudd JHF, van Beek EJR, Tavares A, Virmani R, Berman D, Leipsic JA, Newby DE, Dweck MR. Detection and Prediction of Bioprosthetic Aortic Valve Degeneration. J Am Coll Cardiol. 2019 Mar 19;73(10):1107-1119. doi: 10.1016/j.jacc.2018.12.056. PMID 30871693
- [Derived] Kwiecinski J, Tzolos E, Cartlidge TRG, Fletcher A, Doris MK, Bing R, Tarkin JM, Seidman MA, Gulsin GS, Cruden NL, Barton AK, Uren NG, Williams MC, van Beek EJR, Leipsic J, Dey D, Makkar RR, Slomka PJ, Rudd JHF, Newby DE, Sellers SL, Berman DS, Dweck MR. Native Aortic Valve Disease Progression and Bioprosthetic Valve Degeneration in Patients With Transcatheter Aortic Valve Implantation. Circulation. 2021 Oct 26;144(17):1396-1408. doi: 10.1161/CIRCULATIONAHA.121.056891. Epub 2021 Aug 29. PMID 34455857